CLINICAL TRIAL: NCT00912301
Title: Effect of Chenodeoxycholic Acid on Gastrointestinal Transit and Colonic Functions in Health and Constipation-predominant Irritable Bowel Syndrome (IBS-C)
Brief Title: Cheno Effect on Transit in Health and IBS-C
Acronym: Chenotransit
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Michael Camilleri, M.D., Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-001003; R01DK054681 (NIH); R01DK079866 (NIH); UL1RR024150 (NIH); 1RC1DK086182 (NIH)
Record Dates: First submitted 2009-05-29; First posted 2009-06-03 (Estimated); Results first posted 2012-07-02 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-05

CONDITIONS: Constipation-predominant Irritable Bowel Syndrome
Keywords: chenodeoxycholate, IBS, transit, colon, constipation
MeSH Terms: conditions — Ichthyosis Bullosa of Siemens; Constipation | interventions — Chenodeoxycholic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- NaCDC 500 mg (Experimental): Participants randomized to this arm received 500 mg NaCDC per day for 4 days.
  Interventions: Drug: Sodium chenodeoxycholate (NaCDC)
- NaCDC 1000 mg (Experimental): Participants randomized to this arm received 1000 mg NaCDC per day for 4 days.
  Interventions: Drug: Sodium chenodeoxycholate (NaCDC)
- Placebo (Placebo Comparator): Participants randomized to this arm received a placebo capsule each day for 4 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Sodium chenodeoxycholate (NaCDC) — 500 or 1000 milligrams NaCDC per day each for a period of 4 days
  Other Names: Chenodiol
  Arms: NaCDC 1000 mg; NaCDC 500 mg
Other: Placebo — Placebo capsules with identical appearance to the study drug were prepared by the Mayo Clinic research pharmacy.
  Arms: Placebo

SUMMARY:
The study hypothesis is that the naturally occurring bile acid, chenodeoxycholic acid, induces acceleration of colonic transit in health and in patients with constipation-predominant Irritable Bowel Syndrome (IBS-C).

DETAILED DESCRIPTION:
Hypothesis: A hydrophobic di-alpha hydroxy bile salt, sodium chenodeoxycholate (CDC), delivered in a delayed release capsule to the ileocolonic region of the colon induces acceleration of colonic transit in patients with constipation-predominant IBS.

Methods: We shall study 36 patients with IBS-C, aged 18-65 years, and each treatment group will be balanced on gender and Body Mass Index (BMI) in the randomization. All patients will be assessed for symptoms of functional gastrointestinal disorder or psychological disturbance will be characterized in a standard fashion with questionnaires (Talley et al 1989), the Psychosomatic Symptom Checklist (SCL-90) and the Hospital Anxiety and Depression Inventory [HAD (Zigmond and Snaith 1983)]. With appropriate consent, a venous blood sample will be obtained from each participant for DNA extraction. Fasting Serum 7alpha-hydroxy-4-cholesten-3-one (7alpha-CHO) will be measured in all to ensure they do not have evidence of asymptomatic bile acid malabsorption. The normal range in our lab is <61 ng/mL.

Experimental design: A randomized, double blind, placebo controlled, dose-response parallel group design, with concealed allocation. Participants will undergo an initial baseline colonic transit for 24 hours to obtain Colonic Geometric Center (GC24). Sodium chenodeoxycholate (CDC) will be delivered to the ileocolonic region to assess ascending colon and whole colonic transit in participants with IBS-C; 12 participants per group will be randomized to placebo, 0.5 or 1 gram CDC each for a period of 4 days with the transit study conducted during the last 48 hours of drug ingestion. The CDC will be placed in gelatin capsules that are coated with methacrylate (EUDRAGIT-L®), a pH-sensitive polymer that will result in release of the active ingredient in the terminal ileum.

Experimental procedure: At standardized times (hourly for first 8 hours, and at 12, 24 and 48 h), dual gamma camera scans will be obtained to measure ascending colon and overall colonic transit. Patients will fill daily diaries to evaluate stool, frequency, consistency and ease of passage.

Gastrointestinal and Colonic Transit: A validated scintigraphic method to measure gastric, small bowel, and colonic transit will be used. A methacrylate-coated capsule dissolves in the alkaline pH of the distal ileum to release 111In-labeled activated charcoal particles to evaluate colonic transit on sequential scans. Meanwhile, orally ingested 99 mTc-labeled egg meal allows measurement of gastric and small bowel transit. (Technetium [99mTc] sestamibi (trade name Cardiolite) is a pharmaceutical agent used in nuclear medicine imaging.) We have previously shown that the gastric emptying (GE) at 2 and 4 hours, colonic filling (CF) at 6 hours, and colonic geometric center (GC, weighted average of isotopic counts) in colon at 4, 24 and 48 hours provide excellent summaries of gastric emptying and colonic transit with similar diagnostic accuracy as more detailed, costly, and time-consuming analyses. The normal values for these parameters have been previously published (Cremonini et al).

Scintigraphic gastric emptying and intestinal/colonic transit analysis: A variable region of interest program will be used to measure transit, as in previous studies from our lab. Radioisotope content in each region (gastric, ascending, transverse, descending, rectosigmoid) will be corrected for decay and tissue attenuation or depth.

Anticipated Result: CDC will accelerate whole colonic transit and loosen stool form in patients with constipation predominant IBS.

ELIGIBILITY:
Inclusion Criteria:

Healthy volunteers:

* Age (yr) 18-65
* Gender (F:M)3.5 :1
* Bowel Disease Questionnaire (BDQ) - IBS symptoms negative by Rome III criteria
* Hospital Anxiety/Depression score <8

IBS patients:

* Age (yr) 18-65
* Gender (F:M) 5 :1
* BDQ - IBS symptoms: positive by Rome III criteria
* Hospital Anxiety/Depression score: No restrictions

Exclusion Criteria:

* Abdominal surgery (except appendectomy or cholecystectomy)
* GI medications during the 48h prior to transit measurement
* Aspartate/Alanine transaminases >2 X Upper Limit of Normal (ULN)
* Other Medications except stable doses of estrogen, thyroid, low dose antidepressants of the dopaminergic or serotonergic class

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2009-04; Primary Completion 2009-11 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael L. Camilleri, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Cremonini F, Mullan BP, Camilleri M, Burton DD, Rank MR. Performance characteristics of scintigraphic transit measurements for studies of experimental therapies. Aliment Pharmacol Ther. 2002 Oct;16(10):1781-90. doi: 10.1046/j.1365-2036.2002.01344.x. PMID 12269971
- [Result] Rao AS, Wong BS, Camilleri M, Odunsi-Shiyanbade ST, McKinzie S, Ryks M, Burton D, Carlson P, Lamsam J, Singh R, Zinsmeister AR. Chenodeoxycholate in females with irritable bowel syndrome-constipation: a pharmacodynamic and pharmacogenetic analysis. Gastroenterology. 2010 Nov;139(5):1549-58, 1558.e1. doi: 10.1053/j.gastro.2010.07.052. Epub 2010 Aug 4. PMID 20691689

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled between April 17 and November 20, 2009 from 150 mile geographical area around Mayo Clinic, Rochester, MN.
Pre-assignment Details: 40 patients signed informed consent, but 3 failed screening due to presence of evacuation disorder, and 1 withdrew prior to study due to illness.
Period: Overall Study
Arm/Group | NaCDC 500 mg | NaCDC 1000 mg | Placebo
Started | 11 | 12 | 13
Completed | 11 | 12 | 13
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NaCDC 500 mg | NaCDC 1000 mg | Placebo | Total
Number analyzed (Participants) | 11 | 12 | 13 | 36
Age Continuous [Mean (Standard Deviation); unit: years] | 38.3 (3.3) | 46.1 (2.6) | 40.8 (2.3) | 42 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 12 | 13 | 36
  Male | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 13 | 36

OUTCOME MEASURES:

1. Primary Outcome: Colonic Geometric Center at 24 Hours (GC24)
Description: The scintigraphic method is used to measure colonic transit. An isotope is adsorbed on activated charcoal particles and delivered to the colon in a delayed release capsule. Anterior and posterior gamma images are taken hourly. The geometric center (GC) is the weighted average of counts in the different colonic regions. The scale ranges from 1 to 5; a high GC implies faster colonic transit, a GC of 1 implies all isotope is in the ascending colon, and a GC of 5 implies all isotope is in the stool.
Time Frame: after 4 days of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NaCDC 500 mg | NaCDC 1000 mg | Placebo
Number analyzed (Participants) | 11 | 12 | 13
units on a scale | 3.1 (0.4) | 3.5 (0.4) | 2.2 (0.2)

2. Secondary Outcome: Colonic Transit at 48 Hours (GC48)
Description: as for outcome 1
Time Frame: after 4 days of treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NaCDC 500 mg | NaCDC 1000 mg | Placebo
Number analyzed (Participants) | 11 | 12 | 13
units on a scale | 4.1 (0.3) | 4.3 (0.3) | 3.8 (0.3)

3. Secondary Outcome: Ascending Colon Emptying (AC t_1/2)
Time Frame: after 4 days' treatment
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | NaCDC 500 mg | NaCDC 1000 mg | Placebo
Number analyzed (Participants) | 11 | 12 | 13
hours | 9.5 (2.9) | 8.2 (1.8) | 15.8 (2.5)

4. Secondary Outcome: Stool Consistency
Description: The subjects rated their stool consistency using the Bristol Stool Scale. The Bristol Stool Scale is a medical aid designed to classify the form of human feces into seven categories or types. Types 1 and 2 indicate constipation with 3 and 4 being the "ideal stools" especially the latter, as they are the easiest to defecate, and 5-7 tending towards diarrhea.
Time Frame: after 4 days' treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | NaCDC 500 mg | NaCDC 1000 mg | Placebo
Number analyzed (Participants) | 11 | 12 | 13
units on a scale | 4.4 (0.5) | 4.4 (0.4) | 2.9 (0.3)
Statistical Analysis 1: Comparison: NaCDC 500 mg vs Placebo; Test type: Superiority or Other; p = 0.031, Dunnett's test; pairwise comparison low dose NaCDC against placebo
Statistical Analysis 2: Comparison: NaCDC 1000 mg vs Placebo; Test type: Superiority or Other; p = 0.010, Dunnett's test; pairwise comparison high dose NaCDC against placebo

5. Secondary Outcome: Colonic Filling at 6 Hours
Description: Percent of the radio-labeled meal that reached the colon at 6 hours, indirectly reflecting small bowel transit time.
Time Frame: after 4 days' treatment
Measure: Mean (Standard Deviation); unit: percentage of the radio-labeled meal
Arm/Group | NaCDC 500 mg | NaCDC 1000 mg | Placebo
Number analyzed (Participants) | 11 | 12 | 13
percentage of the radio-labeled meal | 52.6 (6.7) | 54.8 (7.1) | 50.6 (6.7)

ADVERSE EVENTS:
Time Frame: Adverse events were collected during the 4 days of the study.
Arm/Group | NaCDC 500 mg | NaCDC 1000 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 6/11 | 8/12 | 2/13
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NaCDC 500 mg (N=11) | NaCDC 1000 mg (N=12) | Placebo (N=13)
Lower abdominal cramping/pain (Gastrointestinal disorders) | 5 (5) | 5 (5) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Headache (General disorders) | 2 (2) | 2 (2) | 2 (2)
Gas (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0)
Heartburn (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Light-headedness (General disorders) | 1 (1) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No